CLINICAL TRIAL: NCT06014138
Title: Effect of Volatile Sedation on Spontaneous Breathing During Mechanical Ventilation for Patients With the Acute Respiratory Distress Syndrome
Brief Title: Volatile Sedation for Patients With the Acute Respiratory Distress Syndrome
Acronym: ISO-DRIVE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Sedana Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SMRG_318537
Record Dates: First submitted 2023-06-21; First posted 2023-08-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation Complication; Sedation Complication
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Propofol; Isoflurane

STUDY DESIGN:
Intervention Model Description: Prospective, cross-over trial design comparing intravenous versus inhaled volatile sedation
Masking Description: None, open label, physiological study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional intravenous sedation (Active Comparator): Conventional intravenous sedation (e.g. propofol) with short acting opioid, titrated to a clinically prescribed sedation score. Period of observation will be 2 hours pre-cross over and 2 hours post cross over.
  Interventions: Drug: Propofol
- Inhaled volatile sedation (Active Comparator): Inhaled volatile sedation (Isoflurane) delivered via the AnaConDa device for a 6 hour period (2 hours washout of intravenous sedation / wash-in of volatile to achieve stable baseline, followed by 4 hours of observations at steady state) titrated to an equivalent sedation score. During this period opioid infusion should be maintained at baseline level unless clinical indication for titration of dose.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Propofol — Standard care, propofol sedation - 2 hour periods of observation before and after inhaled volatile sedation
  Arms: Conventional intravenous sedation
Drug: Isoflurane — Inhaled volatile sedation for 6 hours - 2 hours wash in / wash out, followed by 4 hours of observations
  Arms: Inhaled volatile sedation

SUMMARY:
This study will investigate how different types of routine sedation may affect patient's breathing whilst on a ventilator in the Intensive Care Unit (ICU). There are different approaches to sedation which may have advantages and disadvantages. During the study patients will receive both intravenous and inhaled volatile sedation (similar to anaesthetic 'gases' used for general anaesthesia) and the drive to breath, breathing efforts and function of the lung will be assessed.

DETAILED DESCRIPTION:
It is routine for patients to be sedated for their comfort and safety whilst on a ventilator in the Intensive Care Unit (ICU). Conventionally sedatives are given intravenously, however inhaled volatile sedation is becoming more popular. Inhaled sedation has recently been approved by the National Institute for Health and Clinical Excellence (NICE) in the United Kingdom (UK).

Whilst being on a ventilator can be life-saving, it can cause potential problems. It is important that the patient interacts well with the ventilator and that their own breathing efforts are well regulated. There is evidence that inhaled sedation can specifically help the lungs when patients have the Acute Respiratory Distress Syndrome (ARDS) and in particular, inhaled sedation does not appear to suppress patient's own breathing as much as conventional sedation. Greater spontaneous breathing by the patient is usually positive but needs to be carefully understood to ensure it is not excessive or damaging to the patient's already injured lungs.

This study of 20 patients is designed to carefully measure the impact of inhaled sedation on the patient's breathing and lung function, in comparison to intravenous sedation. Measurements will be taken whilst on intravenous sedation before the patient is switched to an equivalent level of inhaled sedation for six hours, when the measurements will be repeated. Finally, the patient will go back to their original intravenous sedation and the measurements taken again. This is called a 'cross-over' study and is a good way to evaluate the effect of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Intensive Care Unit (ICU)
* ARDS
* Invasive mechanical ventilation (IMV)
* Spontaneous breathing in pressures support mode (PSV) for less than or equal to 48 hours
* Sedated with intravenous sedation (ie. propofol and / or midazolam and fentanyl or alternate short acting opioid)
* Anticipated to remain on IMV and PSV and with a stable sedation score for a further 24 hours without planned sedation interruption / spontaneous breathing trial or other significant change in the level of ventilator support
* Not receiving / anticipated to receive paralysis
* In supine position

Exclusion Criteria:

* Personal or family history of malignant hyperpyrexia
* Known or suspected elevated intracranial pressure
* High dose vasopressors (ie. Noradrenaline > 0.3mcg/kg/min or equivalent)
* Contra-indication to oesophageal balloon (i.e. oesophageal / upper gastro-intestinal pathology)
* Pregnancy
* High dose oral sedatives (e.g. benzodiazepines) or opioids (e.g. oxycodone / oral morphine) which may affect respiratory drive

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory drive (P0.1) | 8 hours
  Negative pressure in the first 100milliseconds of inspiration (P0.1) - Physiological parameter

SECONDARY OUTCOMES:
Respiratory effort (Pmus) | 8 hours
  End expiratory occlusion pressure (Pmus) - Physiological parameter
Respiratory effort (PMI) | 8 hours
  Pressure Muscle Index (PMI) - Physiological parameter
Respiratory effort (Oesophageal pressure swings) | 8 hours
  Oesophageal pressure swings - Physiological parameter
Gas exchange (PaO2:FiO2 ratio) | 8 hours
  Ratio of arterial partial pressure of oxygen to fractional inspired concentration of oxygen (PaO2:FiO2) - Physiological parameter
Gas exchange (pulmonary shunt fraction (Qs/Qt)) | 8 hours
  Pulmonary shunt fraction (Qs/Qt) - Physiological parameter
Gas exchange ( ratio of ventilatory 'dead space' to tidal volume (Vd/Vt)) | 8 hours
  ratio of ventilatory 'dead space' to tidal volume (Vd/Vt) - Physiological parameter
Gas exchange (volume of carbon dioxide breathed out (VCO2)) | 8 hours
  volume of carbon dioxide breathed out (VCO2) - Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Guy Glover, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No